CLINICAL TRIAL: NCT03344900
Title: Re-Aiming at Hydroxyurea Adherence for Sickle Cell With mHealth
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: University of Memphis (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: REHASH; U01HL133996 (NIH)
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-11

CONDITIONS: Sickle Cell Disease
Keywords: mHealth; Medication adherence; Barriers to adherence
MeSH Terms: conditions — Anemia, Sickle Cell; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase I: It is estimated that 100 participants with SCD will be enrolled for the Phase I portion which will identify barriers to hydroxyurea utilization.
- Phase II: It is estimated that 72 participants with SCD will be enrolled for the Phase II portion of the study which will evaluate the degree of feasibility and acceptance of mHealth intervention on hydroxyurea adherence.

SUMMARY:
National Institutes of Health (NIH)/National Heart, Lung, and Blood Institute (NHLBI) guidelines recommend that hydroxyurea be offered to symptomatic adults and all children with sickle cell disease (SCD) (HbSS and HbSβ0-thal genotypes) age ≥9 months. Research has shown that hydroxyurea reduces hospitalizations and mortality, supporting its effectiveness outside of clinical trials. Hydroxyurea is given as a once-daily oral dose that costs <$1 per day. Despite overwhelming evidence for positive effects, hydroxyurea is vastly underutilized. Given the relative ease of its administration, low cost, and safety profile, barriers to hydroxyurea utilization are primarily constrained to the health system and patient determinants. System-level barriers include insufficient access to SCD-specific care, limited access to medication (due to lack of health coverage), and providers' reluctance in prescribing it; while patient-level barriers include low acceptance (due to insufficient knowledge or misconceptions regarding risks and benefits), and forgetfulness leading to poor adherence.

Mobile health (mHealth) refers to the practice of medicine and public health supported by mobile devices. Short message service (SMS) text messaging (through cell phones) is a widespread means of communication, particularly among adolescents and young adults and is an emerging intervention modality to improve medication adherence. Its low cost, simplicity, and prevalence allow for relatively easy adoption and dissemination in medical practices.

This protocol seeks to examine barriers to hydroxyurea adherence among SCD patients between 15 and 45 years of age who are living in the Memphis region by conducting a needs assessment. In addition to examining these barriers, the needs assessment will provide data that will inform the development of an mHealth application (e.g. mobile phone application) for assisting patients in increasing their medication adherence. The developed mHealth intervention will then undergo a pilot trial to test its acceptability, satisfaction, and feasibility among 56 patients living with SCD.

* To conduct multi-level needs assessment of hydroxyurea utilization barriers and facilitators, in Memphis, Tennessee (Phase I).
* To test the feasibility and acceptance of a patient-informed smart phone application aimed at improving hydroxyurea adherence in the Memphis, Tennessee region, and to estimate the efficacy parameters needed to design a definitive large phase III trial (Phase II).

DETAILED DESCRIPTION:
Data for the needs assessment and pilot trial will be collected from the patients via validated surveys, qualitative methods (e.g., interviews and focus groups), and medical record abstraction.

The study will utilize a Hybrid Effectiveness-Implementation design that will blend both a new intervention to impact the effectiveness of hydroxyurea, text messaging, and study its potential for adoption and dissemination in "real-world" practice settings. In Phase I (formative process evaluation), actionable barriers of hydroxyurea adherence in Memphis, Tennessee, will be identified. The investigators will begin by conducting a broad evaluation of hydroxyurea utilization, impediments and facilitators of hydroxyurea adherence and care management in general for patients with SCD. Next, this information will be merged with patients' preferences for the content of an mHealth intervention, and test it in a local cohort (Phase II). If successful and approved by the Sickle Cell Disease Implementation Consortium (SCDIC) executive committee, this intervention will advance to the next phase, namely, the dissemination and implementation in a larger geographical area (the other SCDIC participating sites in Phase III). We will utilize the RE-AIM framework to evaluate the intervention representativeness and impact during all phases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell disease (any genotype)
* Between the ages of 15 and 44.9 years
* English-speaking

Exclusion Criteria:

* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent

Ages: 15 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will reside in the Memphis, Tennessee, area and meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Compare the number of patients with hydroxyurea barriers or facilitators in hydroxyurea maintenance users and hydroxyurea former users/non-users (Phase I) | From on-study date up to 12 months later
  Multi-level needs assessment of hydroxyurea utilization barriers and facilitators, in Memphis, Tennessee, will be conducted to identify potential factors that affect the barriers or facilitators of hydroxyurea acceptance and that affect the adherence/maintenance of hydroxyurea. Enrollment for Phase I is estimated to be 100. The numbers of patients with barriers or facilitators in hydroxyurea maintenance users and hydroxyurea former users/non-users will be provided and will be compared using Fisher's exact text. This will be done via questionnaires with individuals living with sickle cell disease.
Number of participants who are enrolled and randomized on the study (Phase II) | From study start date through up to 24 months later
  In terms of feasibility of enrollment and randomization, that is, we will assess if we can enroll and randomize 40% (versus an unacceptable rate of 30%) of the approached eligible individuals (56 patients out of 150 approached) in the 24-month accrual duration.
Number of randomized patients completing baseline and 24-week evaluations for both arms | From on-study date up to 24 weeks later
  In terms of the feasibility of conducting a randomized trial, that is, after randomization, per each arm, we will assess if we can have 75% (versus an unacceptable rate of 50%) of randomized individuals (19 patients out of 28 randomized per arm) will complete at least baseline and 24-week evaluations.
Compare the number of participants who report themHealth intervention is useful | Weeks 12 and 24
  Measure the patients' perceived usefulness of mHealth intervention as an aid to hydroxyurea adherence. The proportions of patients who reported the mHealth intervention is useful at weeks 12 and 24 will be provided and will be tested to see if it is significantly different from random at a significance level of 0.05.
The mean and standard deviation of change in satisfaction with mHealth intervention | From on-study date up to 24 weeks
  Measure satisfaction of the intervention by comparing the change in satisfaction measured by the Treatment Satisfaction Questionnaire for Medication (TSQM-9) from baseline to 24 weeks. The change in satisfaction from baseline to 24 weeks will be summarized using mean and standard deviation in the text messaging arm and will be tested using t-test or Wilcoxon signed rank test depending on the normality of the data tested by Shapiro Wilk test at a significance level of 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Jane S. Hankins, MD, MS, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baptist Memorial Hospital, Baptist Clinical Research Institute, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols